CLINICAL TRIAL: NCT00229437
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of Three Doses of TAK-128 in Subjects With Mild to Moderate Diabetic Peripheral Neuropathy
Brief Title: Efficacy and Safety Study of TAK-128 in Treating Subjects With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-04-TL-128-003; U1111-1128-5843 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetic Mononeuropathy; Diabetic Neuralgia; Mononeuropathy, Diabetic; Neuralgia, Diabetic; Diabetic Polyneuropathy; Drug Therapy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- TAK-128 5 mg QD (Experimental)
  Interventions: Drug: TAK-128
- TAK-128 50 mg QD (Experimental)
  Interventions: Drug: TAK-128
- TAK-128 100 mg QD (Experimental)
  Interventions: Drug: TAK-128
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-128 — TAK-128 5 mg, tablets, orally, once daily for up to 6 months.
  Arms: TAK-128 5 mg QD
Drug: TAK-128 — TAK-128 50 mg, tablets, orally, once daily for up to 6 months.
  Arms: TAK-128 50 mg QD
Drug: TAK-128 — TAK-128 100 mg, tablets, orally, once daily for up to 6 months.
  Arms: TAK-128 100 mg QD
Drug: Placebo — TAK-128 placebo-matching tablets, orally, once daily for up to 6 months.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine the efficacy and safety of TAK-128, once daily (QD), in treating subjects with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Polyneuropathy is a frequent complication of diabetes; it affects most individuals after prolonged hyperglycemia, and diabetic neuropathy is very common in the developed world. Chronic, insidious, distal sensorimotor polyneuropathy with autonomic impairment is the most typical form of diabetic neuropathy. Less common, but more florid presentations include autonomic symptoms or painful neuropathy. Although many patients have no or relatively few symptoms, the chronic polyneuropathy and autonomic dysfunction predispose to neurotrophic foot ulceration; consequently, diabetes is the leading cause of amputation today.

Diabetic neuropathy is a dying-back polyneuropathy with distal degeneration of the longest nerve fibers advancing in a centripetal direction. Multiple histopathological changes are observed, but progressive fiber loss is the hallmark of diabetic polyneuropathy. Other important features include endothelial cell basement membrane thickening, segmental demyelination and remyelination, and axonal atrophy. Similar pathological changes are observed in type 1 and type 2 diabetes. The severity of neuropathy as indicated by the stage of nerve fiber loss determines the clinical, electrophysiological, and quantitative sensory threshold features of this disorder. The functional measures of electrophysiological and quantitative sensory thresholds reflect the morphological changes and the clinical features.

Diabetic polyneuropathy is etiologically related to prolonged hyperglycemia with multiple consequences. Although strict glycemic control prevents neuropathy in type 1 patients if maintained for many years, similar interventions in those with type 2 diabetes mellitus are less successful. Type 2 patients may have neuropathy with considerable nerve fiber loss at the time of diagnosis because of unsuspected hyperglycemia in preceding years. Reversal of established neuropathy with strict glycemic control is not certain to occur, even if maintained for many years. Co-morbid disease often interferes with strict management of type 2 diabetes. Even among those with type 1 diabetes, a minority of patients are successful in maintaining prolonged euglycemia.

TAK-128 is a novel synthetic compound being developed as a treatment for diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of childbearing potential must be nonpregnant, nonlactating and on an acceptable form of contraception.
* The subject has fasting clinical laboratory evaluations within the normal reference range for the testing laboratory, or if not, the results must be deemed not clinically significant by the investigator prior to randomization.
* The subject has type 1 or 2 diabetes mellitus using World Health Organization Criteria.
* The subject has mild to moderate peripheral neuropathy defined as:

  * Clinical neuropathy score greater than or equal to 2.5 on the Michigan Neuropathy Screening Instrument.
  * Confirmed abnormality of at least 2 nerve conduction study velocity parameters as defined by the Neurological Core Laboratory.
  * Sural sensory nerve potential amplitude greater than or equal to 1 microvolt.
* The subject's glycosylated hemoglobin is less than or equal to 10%.
* The subject is on stable diabetic therapy for at least 3 months prior to randomization.
* The subject is on stable pain medication for at least 6 weeks prior to randomization, if applicable.
* The subject's creatinine level is less than or equal to 2 mg/dL or 176.8 umol/L.
* The subject is willing to follow an American Diabetes Association or similar recommended dietary regimen.

Exclusion Criteria:

* The subject has a history of other neuropathies due to causes other than diabetes such as alcohol abuse liver or renal disease, uremia, toxic exposure, genetic factors, inflammatory demyelinating diseases, monoclonal gammopathies; or endocrine, metabolic or nutritional disorders (included treated or untreated pernicious anemia).
* The subject has clinical or electrophysiologic evidence of bilateral carpal tunnel syndrome.
* The subject has a significant skin abnormality or ulcerative changes in their lower extremities.
* The subject's body mass index is greater than 40 kg/m2.
* The subject's systolic blood pressure is greater than 160 mm Hg or diastolic blood pressure is greater than 95 mm Hg.
* The subject has a history of myocardial infarction, coronary angioplasty or bypass graft, unstable angina pectoris, transient ischemic attacks, significant electrocardiograms, or documented cerebrovascular accident within 6 months prior to Screening, or is New York Heart Association Functional Cardiac Classification III or IV.
* The subject has an alanine aminotransferase level of greater than 1.5 times the upper limit of normal, active liver disease, or jaundice.
* The subject has a significant, actively treated or unstable pulmonary, gastrointestinal, hepatic, hematologic, musculoskeletal, or endocrine (other than diabetes mellitus or stably treated hypothyroidism) disease.
* The subject has a previous history of cancer, other than basal cell carcinoma, that has not been in remission for at least 5 years prior to the first dose of study drug.
* The subject has taken lipoic acid, linolenic acid (primrose oil), inositol, topiramate, Acetyl-L-Carnitine, nerve growth factors, or capsaicin within 30 days prior to Screening.
* The subject has any other serious disease or condition at Screening or at randomization that might affect life expectancy or make it difficult to successfully manage and follow the subject according to the protocol.
* The subject has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within the past 2 years.
* The subject has a known hypersensitivity to a compound related to TAK-128.
* Subjects can not use any of the following prescription medications throughout the duration of the study, including:

  * Lipoic acid
  * Linolenic acid (primrose oil)
  * Inositol
  * Topiramate
  * Acetyl-L-Carnitine
  * Nerve growth factors
  * Capsaicin
* The subject currently is participating in another investigational study or has participated in an investigational study within the past (30 days or 5 half lives, whichever is longer).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2005-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in composite measure of maximal nerve conduction velocity (Nerve Conduction Studies). | Week 24 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in the electrophysiologic parameters for individual nerves, including amplitudes (Nerve Conduction Studies). | Week 24 or Final Visit
Change from Baseline in vibration perception threshold measurements (Quantitative Sensory Testing). | Weeks 12, 24 or Final Visit
Change from Baseline in pain scores (Short-Form McGill Pain Questionnaire). | Weeks: 8, 12, 16, 20, 24 or Final Visit
Change from Baseline in the neurological examination (Clinical Neurological Examination). | Weeks 12, 24 or Final Visit
Change from Baseline in quality of life index (SF-36 Health Survey). | Weeks: 8, 12, 16, 20, 24 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (48):
- United States (40):
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Huntington Beach, California
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Northridge, California
  - San Francisco, California
  - Torrance, California
  - Tustin, California
  - Aventura, Florida
  - Fort Myers, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Palm Beach Gardens, Florida
  - Plant City, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Flint, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Elizabeth, New Jersey
  - New Brunswick, New Jersey
  - Buffalo, New York
  - Staten Island, New York
  - Greenville, North Carolina
  - Oklahoma City, Oklahoma
  - Morrisville, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Tacoma, Washington
- Canada (8):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Kingston, Ontario
  - North Bay, Ontario
  - Sarina, Ontario
  - Gatineau, Quebec
  - Laval, Quebec
  - Québec, Quebec